CLINICAL TRIAL: NCT00609804
Title: Randomized Phase II Trial of Sorafenib and Erlotinib or Sorafenib Alone in Patients With Advanced Non-Small Cell Lung Cancer Progressing on Erlotinib
Brief Title: Sorafenib and Erlotinib or Sorafenib Alone in Advanced Non-Small Cell Lung Cancer Progressing on Erlotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 162
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Advanced; Erlotinib; Sorafenib; Progressing on erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib+Erlotinib (Experimental): Sorafenib 400 mg twice daily by mouth Erlotinib 150 mg once daily by mouth
  Interventions: Drug: Sorafenib; Drug: Erlotinib
- Sorafenib (Active Comparator): Sorafenib 400 mg twice daily by mouth.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg twice daily by mouth Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
  Other Names: Nexavar
Drug: Erlotinib — Erlotinib 150 mg once daily by mouth
  Other Names: Tarceva
  Arms: Sorafenib+Erlotinib

SUMMARY:
This is a randomized, open-label, multi-center, Phase II study of treatment of patients with advanced NSCLC who have progressed on erlotinib with the combination of sorafenib and erlotinib or sorafenib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage IIIB/IV or relapsed non-small cell lung carcinoma (squamous carcinoma, adenocarcinoma, or large cell carcinoma). Patients with mixed tumors with small-cell elements are ineligible.
2. Patients with no more than 2 prior lines of therapy, with the latest of those therapies being single-agent erlotinib.
3. Evidence of progressive disease on erlotinib as assessed by the treating physician. Erlotinib must be the last treatment for NSCLC prior to enrollment into this study. Patients may be on erlotinib until enrollment. If erlotinib has already been stopped, the period of time off Erlotinib cannot exceed 14 days prior to study enrollment.
4. Patients must have experienced a clinical benefit (complete response [CR], partial response [PR], or stable disease [SD]) from prior therapy with erlotinib for a period of 8 weeks.
5. Patient must have one measurable lesion measuring at least 10 mm in the longest diameter (LD) by spiral computed tomography (CT), or 20 mm with conventional techniques according to the Response Evaluation Criteria in Solid Tumors (RECIST).
6. Recovery from any toxic effects of erlotinib to ≤ grade 1 per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
7. Completion of palliative radiation therapy prior to the start of study treatment. Previously irradiated lesions in the advanced setting cannot be included as target lesions unless clear tumor progression has been observed following the completion of radiation therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
9. Absolute neutrophil count (ANC) >=1,500 and platelets >=75,000 (within 7 days prior to initial study treatment).
10. Hemoglobin >=9 g/dL (within 7 days prior to initial treatment).
11. International normalized ratio (INR) <=1.5 or prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits (WNL) of the institution if not on anticoagulation therapy. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate with the therapeutic range established prior to study treatment initiation.
12. Serum creatinine <=1.5 x institutional upper limit of normal (ULN) within 7 days prior to initial study treatment. If the absolute value is greater than 2mg/dL, the creatinine clearance, calculated according to the Cockroft-Gault formula, must be >=45 mL/min to be eligible.
13. Bilirubin <=1.5 x the ULN; transaminases <=3 x institutional ULN, except in known hepatic metastasis, wherein these may be >=5 x institutional ULN.
14. Patients must be able to understand the nature of this study, give written informed consent, and comply with study requirements.
15. Agreement of male patients (with partners of childbearing potential) and female patients of childbearing potential to use effective contraception to prevent pregnancy during treatment and for a minimum of 90 days thereafter. Additionally, women should not breastfeed during this time.

Exclusion Criteria:

1. Past or current history of neoplasm other than the entry diagnosis, with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone, and a disease-free survival (DFS) >=3 years.
2. Pregnancy or lactation. All females of child-bearing potential must have negative serum or urine pregnancy tests within 7 days prior to study treatment.
3. Prior epithelial growth factor receptor (EGFR) inhibitors, with the exception of erlotinib, are not allowed. This includes both tyrosine kinase inhibitors (TKIs) and monoclonal antibodies. Prior vascular endothelial growth factor (VEGF) inhibitors, with the exception of bevacizumab, are not allowed.
4. Significant cardiac disease within 90 days of starting study treatment including:

   * superior vena cava syndrome
   * new onset angina
   * congestive heart failure (CHF) > Class 2 per New York Heart Association (NYHA) classification
   * arrhythmia
   * valvular heart disease.
5. Myocardial infarction within 6 months prior to initiation of study treatment
6. Cardiomegaly on chest imaging or ventricular hypertrophy on electrocardiogram (ECG) unless the left ventricular ejection fraction (LVEF) is within normal range for the institution.
7. Poorly controlled hypertension (defined as systolic blood pressure [BP] >150 mm Hg and/or diastolic BP >100 mm Hg on antihypertensive medications).
8. Unstable angina (anginal symptoms at rest).
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
10. Presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
11. A serious active infection (> grade 2) at the time of treatment
12. A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
13. Untreated brain metastases. Patients who have treated metastases >=4 weeks out (with surgery and/or radiation therapy) and no evidence of central nervous system (CNS) progression are eligible.
14. Treatment with a non-approved or investigational drug within 28 days of initial study treatment.
15. A major surgical procedure, open biopsy, or significant traumatic injury within 28 days of beginning treatment or anticipation of need for major surgery during the course of the study.
16. Thrombolic or embolic events such as a stroke and transient ischemic attack (TIA) within the past 6 months.
17. Any prior history of hypertensive crisis or hypertensive encephalopathy.
18. Pulmonary hemorrhage/bleeding event >= grade 2 within 28 days of initial study treatment.
19. Any other non-pulmonary hemorrhage/bleeding event >= grade 3 within 28 days of initial study treatment.
20. Evidence or history of bleeding diathesis or coagulopathy.
21. Serious non-healing wound, ulcer, or bone fracture.
22. Use of St. John's Wort or rifampin (rifampicin).
23. Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.
24. Any malabsorption problem.
25. Any condition that impairs the patient's ability to swallow whole pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (16):
- United States (16):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Jackson Oncology Associates, Jackson, Mississippi
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Derived] Spigel DR, Rubin MS, Gian VG, Shipley DL, Burris HA 3rd, Kosloff RA, Shih KC, Quinn R, Greco FA, Hainsworth JD. Sorafenib and continued erlotinib or sorafenib alone in patients with advanced non-small cell lung cancer progressing on erlotinib: A randomized phase II study of the Sarah Cannon Research Institute (SCRI). Lung Cancer. 2017 Nov;113:79-84. doi: 10.1016/j.lungcan.2017.09.007. Epub 2017 Sep 18. PMID 29110854

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib+Erlotinib: Sorafenib 400 mg twice daily by mouth Erlotinib 150 mg once daily by mouth Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
- Sorafenib: Sorafenib: Sorafenib 400 mg twice daily by mouth. Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
Period: Overall Study
Arm/Group | Sorafenib+Erlotinib | Sorafenib
Started | 25 | 28
Completed | 0 (Pts remained on study until required to end treatment due to progression/toxicity/MD decision/etc) | 0 (Pts remained on study until required to end treatment due to progression/toxicity/MD decision/etc)
Not Completed | 25 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib+Erlotinib | Sorafenib | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 83] | 63 [41 to 87] | 65 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Population: All patients on study
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sorafenib+Erlotinib: Sorafenib and Erlotinib: Sorafenib 400 mg twice daily by mouth Erlotinib 150 mg once daily by mouth Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
Arm/Group | Sorafenib+Erlotinib | Sorafenib
Number analyzed (Participants) | 25 | 28
months | 3.1 [1.7 to 3.7] | 1.9 [1.7 to 3.6]

2. Secondary Outcome: Overall Response Rate
Description: The Number of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: All patients on study
Measure: Number; unit: participants
Groups:
- Sorafenib: Sorafenib 400 mg twice daily by mouth. Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
Arm/Group | Sorafenib+Erlotinib | Sorafenib
Number analyzed (Participants) | 25 | 28
participants | 2 | 1

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: Defined as the number of participants with treatment-emergent grade 3/4 adverse events utilizing the National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE) v3.0
Time Frame: 18 months
Population: All patients on study
Measure: Number; unit: participants
Groups:
- Sorafenib and Erlotinib: Sorafenib and Erlotinib: Sorafenib 400 mg twice daily by mouth Erlotinib 150 mg once daily by mouth Study treatment will be given in cycles of 28 days. Patients will be re-staged every 2 treatment cycles (every 8 weeks). Patients with an objective response or stable disease will continue study treatment. Patients will continue until disease progression or intolerable toxicity occurs.
Arm/Group | Sorafenib and Erlotinib | Sorafenib
Number analyzed (Participants) | 25 | 28
participants
  Anemia | 1 | 0
  Fatigue | 4 | 2
  Diarrhea | 4 | 0
  Dehydration | 3 | 2
  Rash/Desquamation | 3 | 2
  Hand-foot skin reaction | 2 | 2
  Dyspnea | 3 | 1
  Hyponatremia | 2 | 3
  Hyperglycemia | 2 | 1
  Lipase increased | 2 | 0
  Anorexia | 1 | 2
  Atrial Fibrillation | 1 | 0
  Cognitive Disturbance | 1 | 0
  Confusion | 1 | 1
  Congestive Heart Failure | 1 | 0
  Constipation | 1 | 1
  Dysphagia | 1 | 0
  Extremity - upper (function) | 1 | 0
  Hypertension | 1 | 1
  Cardiac Ischemia/Infarction | 1 | 0
  Hypokalemia | 1 | 2
  Hypoxia | 1 | 0
  Ileus | 1 | 0
  Infection - Pneumonia | 3 | 0
  Infection - Wound | 1 | 0
  Malaise | 1 | 0
  Nausea | 1 | 2
  Obstruction, GI | 1 | 0
  Pain - abdomen | 1 | 1
  Pain - chest | 2 | 2
  Pain - musculoskeletal | 1 | 8
  Perforation, GI | 1 | 0
  Vomiting | 1 | 1
  Dizziness | 0 | 1
  Infection - urinary tract NOS | 0 | 2
  Neuropathy - cranial | 0 | 1
  Pain - back | 0 | 2
  Pain - head/headache | 0 | 1
  COPD exacerbation | 0 | 1
  Ocular surgery | 0 | 1
  Personality change | 1 | 0
  Respiratory failure | 1 | 0
  Pulmonary embolism | 1 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Sorafenib+Erlotinib | Sorafenib
Serious Adverse Events (participants affected / at risk) | 11/25 | 5/28
Other Adverse Events (participants affected / at risk) | 24/25 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib+Erlotinib (N=25) | Sorafenib (N=28)
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Cardiac disorders - Other, unspecified (Cardiac disorders) | 1 | 0
Cognitive disturbance (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib+Erlotinib (N=25) | Sorafenib (N=28)
Fatigue (General disorders) | 19 | 14
Rash (Skin and subcutaneous tissue disorders) | 17 | 15
Diarrhea (Gastrointestinal disorders) | 15 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Nausea (Gastrointestinal disorders) | 9 | 10
Anorexia (Metabolism and nutrition disorders) | 7 | 10
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 9
Investigations - Other, unknown (Investigations) | 10 | 6
abdominal pain (Gastrointestinal disorders) | 10 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 6
Non-cardiac chest pain (General disorders) | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 6
anemia (Blood and lymphatic system disorders) | 7 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Alkaline phosphatase increased (Investigations) | 3 | 7
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 4 | 6
Creatinine increased (Investigations) | 5 | 5
Platelet count decreased (Investigations) | 6 | 4
Vomiting (Gastrointestinal disorders) | 7 | 3
Weight loss (Investigations) | 6 | 4
White blood cell decreased (Investigations) | 5 | 5
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 3
Hypertension (Vascular disorders) | 4 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 4
Headache (Nervous system disorders) | 2 | 5
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 5 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Fever (General disorders) | 1 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4
Mucositis (Gastrointestinal disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2
Lipase increased (Investigations) | 3 | 1
Respiratory, thoracic and mediastinal disorders - Other, unknown (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Serum amylase increased (Investigations) | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Bronchial infection (Infections and infestations) | 2 | 1
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 1 | 2
Chills (General disorders) | 1 | 2
Confusion (Psychiatric disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
dyspepsia (Gastrointestinal disorders) | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Infections and infestations - Other, pneumonia (Infections and infestations) | 2 | 1
Investigations - Other, blood urea nitrogen increased (Investigations) | 1 | 2
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nervous system disorders - Other, unknown (Nervous system disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders - Other, hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 1
Skin and subcutaneous tissue disorders - Other, skin changes (Skin and subcutaneous tissue disorders) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites